CLINICAL TRIAL: NCT06692114
Title: A Preliminary Study on the Efficacy and Influencing Factors of Deep Transcranial Magnetic Stimulation in the Treatment of Obsessive-compulsive Disorder
Brief Title: Efficacy and Influencing Factors of Deep Transcranial Magnetic Stimulation in the Treatment of OCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhen Wang (Other)
Responsible Party: Sponsor-Investigator, Zhen Wang, vice-president, Shanghai Mental Health Center
Organization: Shanghai Mental Health Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMHC-OCD-012
Record Dates: First submitted 2024-08-30; First posted 2024-11-18 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: deep transcranial magnetic stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active treatment group (Experimental): The resting motor threshold (RMT) of the patient was measured before the first treatment. Symptom induction was performed before each treatment to achieve moderate anxiety in patients. The magnetic stimulation intensity was 100% RMT, using the deep transcranial magnetic stimulation coil H7 for treatment, with the stimulation area being the anterior cingulate cortex (ACC) and medial prefrontal cortex (mPFC). Treatment was administered twice daily for 20 minutes each time for 2 weeks.
  Interventions: Device: Deep Transcranial Magnetic Stimulation, DTMS active
- sham group (Sham Comparator): The same RMT test as the active treatment group was accepted, and symptom induction was performed before treatment to achieve moderate anxiety. During treatment, the coil in the shame treatment group only produces sound and scalp vibration, and does not generate a real magnetic field. There is no other difference between the two coils. The frequency and number of treatments were the same as those in the active treatment group.
  Interventions: Device: Deep Transcranial Magnetic Stimulation, DTMS sham

INTERVENTIONS:
Device: Deep Transcranial Magnetic Stimulation, DTMS active — The treatment plan is to perform 2 treatments per day for 20 minutes each time, for a total of 28 treatments. Each treatment stimulates at a frequency of 20 Hz for 2 seconds, with a sequence interval of 20 seconds. Each treatment consists of 50 sequences, for a total of 2000 pulses.
  Arms: active treatment group
Device: Deep Transcranial Magnetic Stimulation, DTMS sham — The treatment plan is to perform 2 treatments per day for 20 minutes each time, for a total of 28 treatments. Compared with active treatment, the sham stimulation coil only produced sound and scalp vibration.
  Arms: sham group

SUMMARY:
This study aims to explore the efficacy and influencing of accelerated dTMS (deep Transcranial Magnetic Stimulation) treatment in patients with obsessive-compulsive disorder (OCD), and explores the potential neural mechanisms of treatment effect by magnetic resonance imaging (MRI) and electroencephalography (EEG).

DETAILED DESCRIPTION:
The study is to recruit eligible patients with obsessive-compulsive disorder (OCD) from the Shanghai Mental Health Center for deep transcranial magnetic stimulation (dTMS) intervention, and recruit healthy controls who meet the enrollment criteria from the community. Among them, patients with OCD will be randomly divided into a real stimulation group and a sham stimulation group. After baseline assessment, dTMS treatment will be administered twice a day. EEG data collection, MRI data, cognitive tasks, psychological self-assessment scales and clinical symptom assessment will be conducted before treatment and 2 weeks after treatment. During the treatment process, patients will receive two treatments per day, each lasting 20 minutes, for a total of 2 weeks, or 28 treatments in total.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 50, both genders are welcome.
* DSM-5 criteria for OCD.
* Y-BOCS total score ≥ 20 despite therapeutic-dose SRI treatment or completion of at least one full course of CBT. The treatment regimen must have been stable for at least 8 weeks prior to enrollment and remain unchanged throughout the study.
* More than 9 years of education.
* Right-handed.

Exclusion Criteria:

* Any additional current psychiatric comorbidity, except for obsessive- compulsive personality disorder.
* Severe obsessive symptoms prevent the completion of necessary assessments.
* Has a history of receiving ECT therapy.
* Has received rTMS or tDCS treatment within the past two months.
* Has severe physical illnesses or any physical conditions that can induce epilepsy or intracranial hypertension, including cardiovascular and respiratory diseases, among others.
* Has a past history of neurological disorders (such as epilepsy, cerebrovascular accidents, etc.) or brain injuries, or a history of brain surgery.
* Has implanted medical devices such as intracranial stents, cardiac pacemakers, coronary stents, cochlear implants, etc.
* Serious suicide risk.
* Pregnancy or nursing of an infant.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
To explore the differences in treatment efficacy between active and sham dTMS in patients with OCD | baseline,2weeks,4weeks
  It assesses the severity of OCD symptoms. The Y-BOCS scale ranges from 0 to 40, with 0 being no symptoms and 40 being severe.
  The primary outcome measure percent reduction of Y-BOCS scores at completion of the dTMS treatment.

SECONDARY OUTCOMES:
To explore the differences in treatment efficacy between active and sham dTMS in patients with OCD | baseline,2 weeks, 4 weeks
  The secondary outcome measure was the response rate to the treatment, which was defined as a reduction of at least 35% in Yale-Brown Obsessive Compulsive Scale (Y-BOCS)
Change in The Beck Depression Inventory (BDI) | baseline,2 weeks, 4 weeks
  It is a 21-item self-report measure scored on a 4-point Likert-type scale to summarize recent symptoms of depression.
Change in the The Beck Anxiety Inventory (BAI) | baseline,2 weeks, 4 weeks
  It is a 21-item self-report inventory that is used for measuring the severity of anxiety

OTHER OUTCOMES:
Attention Network Task (ANT) | Up to 2 weeks
  Have patients allocate their attention and process information through tasks processed by a grid structure. Monitor whether there are any changes in patients' attention after treatment.
Rapid Serial Visual Presentation (RSVP) | Up to 2 weeks
  Use programs to rapidly present image stimuli in order to assess patients' attention, recognition, or judgment abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Wang, PhD，MD, Principal Investigator — Study Principal Investigato
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China